CLINICAL TRIAL: NCT06927310
Title: A Multicenter, Randomized, Open-Label, Active-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Inpegsomatropin Injection, s.c Once a Week, Compared With Recombinant Human Growth Hormone (rhGH) Injection in Children With Idiopathic Short Stature (ISS).
Brief Title: The Efficacy and Safety of Inpegsomatropin Injection in Children With Idiopathic Short Stature
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGPESEN-4-2-001
Record Dates: First submitted 2025-04-06; First posted 2025-04-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Short Stature
Keywords: Inpegsomatropin Injection; Recombinant Human Growth Hormone Injection
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpegsomatropin group (Experimental)
  Interventions: Drug: Inpegsomatropin Injection
- rhGH group (Active Comparator)
  Interventions: Drug: Recombinant Human Growth Hormone Injection

INTERVENTIONS:
Drug: Inpegsomatropin Injection — Inpegsomatropin injection, 280 μg/kg/week, s.c., once weekly, for 52 consecutive weeks.
  Arms: Inpegsomatropin group
Drug: Recombinant Human Growth Hormone Injection — Recombinant Human Growth Hormone Injection, 350 μg/kg/week, s.c., divided into 7 doses, i.e., 50 μg/kg/day (0.15 IU/kg/day), once daily for 52 consecutive weeks.
  Arms: rhGH group

SUMMARY:
This is a multicenter, randomized, open-label, active-controlled Phase III clinical trial to evaluate the efficacy and safety of Inpegsomatropin injection，once a week，compared with recombinant human growth hormone (rhGH) in children with idiopathic short stature (ISS). It plans to enroll 300 children with ISS, who will be randomized , stratified by gender and age, and assigned to either the experimental group or the positive controlled group. Each participant will undergo a screening period (up to 12 weeks), a treatment period (52 weeks), and a post-treatment follow-up period (5 weeks). And the safety and efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal children: boys aged ≥3 years and <11 years at screening with testicular volume <4 mL; girls aged ≥3 years and <10 years at screening with breast development at Tanner Stage I, i.e., no palpable breast glandular tissue.
* Compared to chronological age, bone age is advanced by no more than 1 year or delayed by no more than 2 years (i.e., -2 years ≤ bone age - chronological age ≤ 1 year).
* Height at screening is below -2 standard deviations (SD) from the mean for age and sex, with height reference to Appendix 1.
* Body mass index (BMI) is within the 5th to 95th percentile for age and sex of healthy children, with reference to Appendix 2.
* Peak GH level ≥10.0 ng/ml in at least one GH stimulation test.
* No prior systemic pharmacological treatment for growth promotion (continuous use ≥1 month), including but not limited to growth hormone, insulin-like growth factor 1 (IGF-1), etc.
* The legal guardian understands and signs the informed consent form. If the participants is ≥8 years old, they must also sign the informed consent form. For participants under 8 years old who are able to express their consent, their assent should be clearly documented.

Exclusion Criteria:

* Individuals with closed epiphyses;
* Other types of growth and developmental abnormalities, including confirmed or highly suspected growth hormone deficiency (GHD), Noonan syndrome, Prader-Willi syndrome, Russell-Silver syndrome, Turner syndrome, small for gestational age, short stature due to SHOX gene abnormalities, growth delay due to malnutrition, growth delay due to hypothyroidism, and other short statures with a clear etiology; genetic testing results must be obtained before randomization to exclude short stature caused by definite genetic abnormalities;
* Individuals who have participated in any other clinical trial within 3 months prior to screening and have received pharmacological or non-pharmacological interventions;
* Individuals who received inhaled corticosteroids for more than 2 consecutive weeks, or oral or intravenous corticosteroids for more than 1 consecutive week, within the 3 months prior to screening;
* Individuals who are currently receiving or require long-term treatment with other therapies that may affect growth, including but not limited to methylphenidate, sex hormones, gonadotropin-releasing hormone analogs, aromatase inhibitors, anabolic agents, insulin, etc.;
* Individuals with abnormal liver or kidney function at screening (ALT > 1.5 times the upper limit of normal, Cr > upper limit of normal);
* Individuals diagnosed with diabetes mellitus, or with fasting blood glucose ≥6.1 mmol/L on two consecutive occasions;
* Individuals with chronic infectious diseases, such as chronic hepatitis B;
* Individuals with systemic chronic diseases, such as moderate to severe anemia, malnutrition, hypothyroidism, chronic kidney disease, cardiovascular diseases (e.g., dilated cardiomyopathy, etc.), psychiatric and psychological disorders, or those with congenital anomalies requiring clinical intervention as determined by the investigator;
* Individuals with congenital skeletal abnormalities, or those with scoliosis exceeding 15°, limping, or a history of slipped capital femoral epiphysis;
* Individuals with a history of increased intracranial pressure;
* Individuals with a history of malignancy or currently having active malignancy, including intracranial tumors;
* Individuals with severe allergic constitutions, or known allergies to growth hormone or its excipients;
* Individuals with any other disease that the investigator deems may endanger the subject's safety or compromise compliance with the study protocol.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Growth velocity (HV, cm/year). | Week 52

SECONDARY OUTCOMES:
Change in height standard deviation score from baseline (△HT SDS) | From baseline to all follow-up time points at Week 52
Change in growth velocity from baseline (△HV) | From baseline to all follow-up time points at Week 52
Change in insulin-like growth factor 1 standard deviation score from baseline (△IGF-1 SDS) | From baseline to all follow-up time points at Week 52
The ratio of the change in bone age to the change in chronological age (△BA/△CA) | From baseline to all follow-up time points at Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Ph.D, Principal Investigator — Tongji Hospital
Locations (38):
- China (38):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Capital Institute of Pediatrics, Beijing (SHOUER), Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Maternity and Child Care Hospital, Lanzhou, Gansu
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Wuhan Children's Hospital, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital Affiliated to Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - The Affiliated Women's and Children's Hospital of Ningbo University, Ningbo, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Sanya Central Hospital, Hainan
  - Hangzhou First People's Hospital, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The First Affiliated Hospital of Henan University of Science and Technology, Henan
  - Jiaxing First Hospital, Jiaxing
  - Affiliated Hospital of Jining Medical University, Jining
  - Kunming Children's Hospital, Kunming
  - Nanjing Children's Hospital, Nanjing
  - Qingdao Women and Children's Hospital, Qingdao
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Renmin Hospital of Wuhan University, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang
  - Yuncheng Central Hospital, Yuncheng
  - Zhuzhou Central Hospital, Zhuzhou

IPD SHARING:
Plan to Share IPD: No